CLINICAL TRIAL: NCT05436665
Title: The Belgian Endothelial Surgical Transplant of the Cornea:Clinical and Patient-reported Outcomes of Descemet Stripping Automated Endothelial Keratoplasty(DSAEK) Versus Descemet Membrane Endothelial Keratoplasty(DMEK)
Brief Title: The Belgian Endothelial Surgical Transplant of the Cornea
Acronym: BESTCornea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UZAntwerpen
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Corneal Edema; Corneal Endothelial Disorder; Fuchs' Endothelial Dystrophy; Bullous Keratopathy; Pseudophakic Bullous Keratopathy
Keywords: DMEK; DSAEK; UT-DSAEK
MeSH Terms: conditions — Corneal Edema; Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Intervention Model Description: After the patient has been screened and deemed eligible for participation, and the informed consent of the patient has been obtained, the patients will be included in the study. Once the inclusion data is entered by a member of the study personnel into the trial software, allocation of the patient to a treatment arm will take place using minimisation.
  The allocation will be performed with an equal 1:1 allocation to DSAEK or DMEK with minimisation using the following stratification of participant factors:
  * Surgical Indication (i.e., Fuchs' endothelial dystrophy and non Fuch's endothelial dystrophy);
  * Surgical site;
  * Preoperative visual acuity (Patients with 0.6 LogMAR BCVA or lower (i.e., better vision) and patients with LogMAR BCVA higher than 0.6 LogMAR (i.e., worse vision).
  The minimisation will be performed by the study team using the online allocation software QMinim.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, the treating surgeons will be unblinded to the graft type. The outcomes will be assess by a blinded assessor and the quality of life questionnaires will be completed by the patient themselves, with assistance from the blinded assessor as needed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-thin Descemet Stripping Automated Endothelial Keratoplasty (UT-DSAEK) (Active Comparator): Ultra-thin Descemet Stripping Automated Endothelial Keratoplasty (UT-DSAEK) refers to the use of a corneal endothelial/Descemet graft with a thin layer of stroma (<110um) attached.
  The cornea is made up of 5 layers, all of which work to provide a clear image on the retina. The innermost layer of cells, the endothelium, is responsible for pumping fluid out of the cornea and keeping it transparent: a normal endothelium is essential to keeping the cornea clear. The endothelium lies on a membrane called the Descemet membrane. The thickest layer of the cornea is called the stroma and this provides rigidity and strength to the cornea. When the corneal endothelium fails, it cannot regrow and the best treatment is to replace the cells with healthy donor cells. This is called a corneal endothelial transplantation or endothelial keratoplasty.
  In the DSAEK technique, a piece of the donor's endothelium is transplanted with a supporting layer of donor stroma.
  Interventions: Procedure: UT-DSAEK
- Descemet membrane endothelial keratoplasty (DMEK) (Active Comparator): Descemet membrane endothelial keratoplasty refers to the use of a corneal endothelial/Descemet graft with no layer of associated stroma (15-20um thick).
  The cornea is made up of 5 layers, all of which work to provide a clear image on the retina. The innermost layer of cells, the endothelium, is responsible for pumping fluid out of the cornea and keeping it transparent: a normal endothelium is essential to keeping the cornea clear. The endothelium lies on a membrane called the Descemet membrane. The thickest layer of the cornea is called the stroma and this provides rigidity and strength to the cornea. When the corneal endothelium fails, it cannot regrow and the best treatment is to replace the cells with healthy donor cells. This is called a corneal endothelial transplantation or endothelial keratoplasty.
  In the DMEK technique only a piece of donor endothelium layer is together with its supporting membrane (the Descemet membrane), is transplanted.
  Interventions: Procedure: DMEK

INTERVENTIONS:
Procedure: UT-DSAEK — The main incision (3.5-5mm) is created at the corneal limbus or via a cornea-scleral tunnel with 2-3 smaller (approx. 1mm) paracentesis incisions. An ophthalmic viscosurgical device (OVD) or a continuous infusion of water or air can be used to maintain the stability of the anterior chamber, according to the surgeon's preference. The corneal endothelium is scored using a scoring instrument and the central diseased corneal endothelium is removed. Once the anterior chamber is prepared, OVD or air has been removed, then the eye is ready for the new corneal graft.
  The pre-cut corneal tissue delivered by the bank is then gently rinsed and may be stained with 0.06% trypan blue if required. The tissue is loaded into a glide or injector, and pulled into the anterior chamber using a smooth-tipped micro-forceps (e.g., Busin forceps). Once the graft enters the eye, it is lifted to the posterior cornea. The graft is further centred using air (or SF6 Gas) in the anterior chamber.
  Other Names: Ultra-Thin Descemet Stripping Automated Endothelial Keratoplasty
  Arms: Ultra-thin Descemet Stripping Automated Endothelial Keratoplasty (UT-DSAEK)
Procedure: DMEK — The main incision (2.8-3mm) is created superior or temporally at the corneal limbus and is accompanied by 2-3 smaller paracentesis incisions. An ophthalmic viscosurgical device (OVD) or a continuous infusion of water or air can be used to maintain the stability of the anterior chamber. The corneal endothelium is scored using a scoring instrument and the central diseased corneal endothelium is removed.
  The DMEK roll is poured into a basin and rinsed. The graft is then stained with 0.06% trypan blue to aid in graft visualization. The graft is loaded into an injector and introduced into the anterior chamber. The graft is unrolled using external manoeuvres and once unrolled, it is lifted to the back of the cornea. The eye is then pressurised with a full air fill from 10 to 120 minutes. The pressure is then reduced and the case is completed by suturing any incisions required.
  Other Names: Descemet Membrane Endothelial Keratoplasty
  Arms: Descemet membrane endothelial keratoplasty (DMEK)

SUMMARY:
This study is designed as a randomised multicentric parallel group pragmatic trial of Descemet Stripping Automated Endothelial Keratoplasty (DSAEK) versus Descemet Membrane Endothelial Keratoplasty (DMEK) in corneal endothelial decompensation. the purpose is to compare the clinical and patient reported outcomes of both therapies across a broad range of indications.

DETAILED DESCRIPTION:
The current problem concerns variability in the provision of corneal endothelial keratoplasties available to patients in Belgium. Some patients receive DSAEK and some (albeit fewer) receive DMEK. Currently the type of corneal graft that a patient receives depends on the treating surgeon opinions.

In this study 220 patients in 11 surgical centres will be recruited and allocated to one of the two surgical options. Both the Ultrathin DSAEK and DMEK grafts will be prepared by corneal banks in the University Hospital of Liege and University Hospital of Antwerp respectively. Patients will be examined preoperatively and postoperatively at 3, 6 and 12 months. Clinical information such as best-corrected visual acuity and refraction will be collected as well as quality of life information based on the EQ-5D-5L and the VFQ 25 assessment tools. These data be used to compare the interventions both on the clinical level as well as from the patient perspective.

ELIGIBILITY:
Inclusion Criteria:

* Fuchs Endothelial Dystrophy (FED);
* Bullous Keratopathy (BK);
* Other miscellaneous causes of endothelial dysfunction including decompensation of a previous corneal graft;
* Pseudophakic (post cataract surgery);
* Patients over 18 with the capacity to read and to understand the study information and to give informed consent, as well as study quality of life questionnaires;
* Patients willing and capable to attend the 3, 6, and 12-month follow-up appointments.

Exclusion Criteria:

* Inability to provide informed consent;
* Patients unable to attend the proposed follow up;
* Inclusion of the fellow eye in the study;
* Complex surgery combined with multiple pathologies (i.e., glaucoma surgery);
* Other contraindications to lamellar corneas surgery;
* Patients who elect not to participate;
* Patients under 18 years of age;
* Patients that are currently pregnant or breastfeeding;
* Phakic patients with no direct plan to perform cataract surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
BCVA 12m | 12 months
  Best-corrected visual acuity expressed in LogMAR

SECONDARY OUTCOMES:
BCVA 3 and 6m | 3 and 6 months
  Best-corrected visual acuity expressed in LogMAR
UCVA 3,6 and12m | 3, 6 and 12 months
  Uncorrected visual acuity expressed in LogMAR
Change in refraction | 3, 6 and 12 months
  Change in objective refraction - spectacle correction
Proportion of high vision | 12 months
  Proportion of patients to achieve 0.2 LogMAR visual acuity or less
EQ-5D-5L | 3, 6 and 12 months
  Quality of life measured by the fifth level EuroQol (EQ-5L) instrument where five dimensions are scored at 5 levels - the higher the level, the worse the health state. The digits for the five dimensions can be combined to a 5-digit number to describe the patient's health state
VFQ 25 | 3, 6 and 12 months
  Vision related quality of life measured by the Visual Function Questionnaire(VFQ-25) scored on a scale of 0-100, with a higher score reporesenting higher quality of vision related quality of life.
ECC | 3, 6 and 12 months
  Endothelial cell count
CCT | 3, 6 and 12 months
  Central corneal thickness
Complications | 12 months
  Complications associated with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sorcha Ni Dhubhghaill, MBBCh, PhD, Study Director — Universitair Ziekenhuis Brussel; Carina Koppen, MD, PhD, Study Chair — University Hospital, Antwerp; Bernard Duchesne, MD, PhD, Study Chair — University Hospital Liege
Locations (11):
- Belgium (11):
  - Antwerp University Hospital, Edegem, Antwerp
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - AZ Sint-Jan Brugge, Bruges, West-Vlaanderen
  - AZ Imelda, Bonheiden
  - Erasmus ziekenhuis Brussel, Brussels
  - UZ Brussel, Brussels
  - AZ Monica (campus Deurne), Deurne
  - Ziekenhuis Oost-Limburg (ZOL), Genk
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHU Liège, Liège

IPD SHARING:
Plan to Share IPD: Yes
Data sharing of the final trial dataset will be offered in the following manner:
  The Chief Investigator, Trial Steering Committee, and the Sponsor (including data monitors) will have access to the trial dataset, but a site's Prinicpal Investigator may submit a request for data access.
  This will be discussed and approved by the Trial Steering Committee. Upon conclusion of the trial, individual participant data that underlie the results reported in the article (after deidentification) will be shared upon the request of any relevant interested party.
  Access to the final trial dataset by other parties: reasonable requests for access to trial data from other parties will be considered and approved in writing where appropriate, following formal application to the Trial Steering Committee (bestcornea@uza.be).
Supporting Information: Study Protocol
Time Frame: The article with regards to the study protocol is now under revision in an open acces medical journal.
Access Criteria: The article with regards to the study protocol will be published in an open access medical journal.

REFERENCES:
- [Derived] de Bruyn B, Ni Dhubhghaill S, Claerhout I, Claes K, Deconinck A, Delbeke H, Huizing M, Krolo I, Muijzer M, Oellerich S, Roels D, Termote K, Van den Bogerd B, Van Gerwen V, Verhaegen I, Wisse R, Wouters K, Consortium TBC, Duchesne B, Koppen C. Belgian Endothelial Surgical Transplant of the Cornea (BEST cornea) protocol: clinical and patient-reported outcomes of Ultra-Thin Descemet Stripping Automated Endothelial Keratoplasty (UT-DSAEK) versus Descemet Membrane Endothelial Keratoplasty (DMEK) - a multicentric, randomised, parallel group pragmatic trial in corneal endothelial decompensation. BMJ Open. 2023 Sep 15;13(9):e072333. doi: 10.1136/bmjopen-2023-072333. PMID 37714670